CLINICAL TRIAL: NCT00746109
Title: Randomized Clinical Trial of Wound Packing Following Incision and Drainage of Superficial Skin Abscesses in the Pediatric Emergency Department
Brief Title: Study of Wound Packing After Superficial Skin Abscess Drainage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Michael Mojica, New York University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-143
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2011-01

CONDITIONS: Abscess; Skin Diseases, Infectious; Boils; Furuncle; Carbuncle; Folliculitis; Cellulitis; Wounds
Keywords: randomized; clinical trial; ultrasound; prospective; abscess; packing; incision and drainage; superficial soft tissue infection
MeSH Terms: conditions — Abscess; Skin Diseases, Infectious; Furunculosis; Carbuncle; Folliculitis; Cellulitis; Wounds and Injuries; Surgical Wound

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NOPACKING (Placebo Comparator): The comparison group will undergo a routine incision and drainage procedure but will not have packing placed inside the abscess cavity.
  Interventions: Procedure: NoPacking
- PACKING (Experimental): This group will receive wound packing as per usual protocol
  Interventions: Procedure: Wound packing

INTERVENTIONS:
Procedure: Wound packing — 1/4" non-iodoform packing loosely placed inside abscess cavity.
  Arms: PACKING
Procedure: NoPacking — This is a routine incision and drainage procedure but without the use of packing. Sterile gauze dressing will be placed over the abscess cavity.
  Arms: NOPACKING

SUMMARY:
Superficial skin and soft tissue abscess are frequently managed by opening them up with a procedure called "incision and drainage". It is routine practice in the United States to place packing material inside the abscess cavity after opening them up, in order to promote better wound healing and limit abscess recurrence. However, this practice has never been systematically studied or proven to decrease complications or improve healing. Patients with wound packing usually return to the emergency room or practice setting for multiple "wound checks" and dressing/packing changes which lead to missed days from work or school and utilization of healthcare resources. This procedure can often be painful and may even require conscious sedation (and the risks entailed) especially in children. With rates of superficial skin and soft tissue abscesses on the rise, and emergency room resources being stretched, it is important to determine whether packing wounds is necessary or even advantageous to patients.

This study is the first to systematically evaluate the efficacy of wound packing after superficial skin or soft tissue abscess incision and drainage in children. The investigators will be evaluating wound healing, complications, recurrence and pain associated with packing both short and long term. In addition, the investigators will also be evaluating the utility of bedside point-of-care ultrasound use in predicting the presence of pus inside the abscess cavity. This test may be useful to determine whether incision and drainage is necessary for an individual who has a skin infection that is suspicious for an abscess.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 - 24 years (i.e. any child seen in PED)
* Suspected abscess deemed to need incision & drainage by attending physician or fellow
* Size of abscess is greater than or equal to 1cm
* Parent or patient consent, and child assent

Exclusion Criteria:

* Location of abscess on face, perianal, or genitals
* History of recurrent or chronic abscess
* Multiple abscesses requiring drainage at current visit
* Immunocompromised or unstable patient
* HIV, transplant recipient, immune deficiency syndrome
* immunosuppressive medications
* Wound already open/draining
* Previous participation in trial
* Patient will not be following up / managed by PES (e.g. surgical site)

Ages: 1 Year to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Healing (resolution, cosmesis, complications and recurrence) | one month
Ultrasound test characteristics | day one

SECONDARY OUTCOMES:
Parental/patient satisfaction | one month
Cost-effectiveness | one month

CONTACTS AND LOCATIONS:
Locations (1):
- New York University / Bellevue Hospital Center, New York, New York, United States

REFERENCES:
- [Derived] Kessler DO, Krantz A, Mojica M. Randomized trial comparing wound packing to no wound packing following incision and drainage of superficial skin abscesses in the pediatric emergency department. Pediatr Emerg Care. 2012 Jun;28(6):514-7. doi: 10.1097/PEC.0b013e3182587b20. PMID 22653459